CLINICAL TRIAL: NCT04593160
Title: Efficacy of Preoperative Diclofenac Potassium- Acetaminophen Combination on Anesthetic Success in Patients With Symptomatic Irreversible Pulpitis: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sovana Tarek, Postgraduate student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CU-ENDO-6-10-2020.
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Symptomatic Irreversible Pulpitis
MeSH Terms: interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diclofenac potassium- acetaminophen combination (Experimental): Preoperative single dose of diclofenac potassium(50mg)- acetaminophen(1000mg) combination
  Interventions: Drug: Diclofenac potassium- acetaminophen combination
- Diclofenac potassium (Experimental): Preoperative single dose of diclofenac potassium(50mg)
  Interventions: Drug: Diclofenac potassium
- Placebo (Placebo Comparator): Preoperative single dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac potassium- acetaminophen combination — Preoperative single dose of diclofenac potassium(50mg)- acetaminophen(1000mg) combination
  Arms: Diclofenac potassium- acetaminophen combination
Drug: Diclofenac potassium — Preoperative single dose of diclofenac potassium(50mg)
  Arms: Diclofenac potassium
Drug: Placebo — Preoperative single dose of placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of preoperative a single-dose of 50 mg diclofenac potassium- 1000mg acetaminophen combination compared to diclofenac potassium alone or placebo on local anesthetic success and postoperative pain in patients with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
Patients with moderate-to-severe preoperative pain are selected. Patients receive either a single-dose of diclofenac potassium (50mg)- acetaminophen (1000mg) combination, diclofenac potassium (50mg) alone or a placebo tablet as a control. All patients will receive the assigned premedication one hour before single-visit root canal treatment. Anesthetic success of inferior alveolar nerve block will be assessed during access and instrumentation. Postoperative endodontic pain is measured at the following time points: 6,12,24,48,72h and 7 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic irreversible pulpitis with/without mechanical allodynia
* Patients with moderato to severe spontaneous pain
* Mandibular molars
* Patients with the ability to understand and use the pain scale
* Patients accepting enrollment in the study

Exclusion Criteria:

* Patients allergic to any medication or material to be used in the study
* Pregnant and lactating females
* Patients taking medications affecting pain perception in the last 12 hours
* Patients having more than one symptomatic molar in the same quadrant
* Patients with contributory medical history (ASA > II)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Anesthetic success of inferior alveolar nerve block | During the treatment
  Will be recorded by 11 point NRS consisting of numbers from 0 through 10. 0: reading represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain" 0: reading represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain". Success will be defined as no to mild pain.

SECONDARY OUTCOMES:
Postoperative pain at 6 hours | 6 hours
  Will be recorded by 11 point NRS consisting of numbers from 0 through 10. 0: reading represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain" 0: reading represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain"
Postoperative pain at 12 hours | 12 hours
  Will be recorded by 11 point NRS consisting of numbers from 0 through 10. 0: reading represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain" 0: reading represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain"
Postoperative pain at 24 hours | 24 hours
  represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain" 0: reading represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain"
Postoperative pain at 48 hours | 48 hours
  represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain" 0: reading represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain"
Postoperative pain at 72 hours | 72 hours
  represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain" 0: reading represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain"
Postoperative pain at 7 days | 7 days
  represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain" 0: reading represents "no pain" 1-3 : readings represent "mild pain" 4-6 : readings represent "moderate pain" 7-10 : readings represent "severe pain"

REFERENCES:
- [Background] Nagendrababu V, Pulikkotil SJ, Veettil SK, Teerawattanapong N, Setzer FC. Effect of Nonsteroidal Anti-inflammatory Drug as an Oral Premedication on the Anesthetic Success of Inferior Alveolar Nerve Block in Treatment of Irreversible Pulpitis: A Systematic Review with Meta-analysis and Trial Sequential Analysis. J Endod. 2018 Jun;44(6):914-922.e2. doi: 10.1016/j.joen.2018.02.017. Epub 2018 Apr 27. PMID 29709297
- [Background] Ianiro SR, Jeansonne BG, McNeal SF, Eleazer PD. The effect of preoperative acetaminophen or a combination of acetaminophen and Ibuprofen on the success of inferior alveolar nerve block for teeth with irreversible pulpitis. J Endod. 2007 Jan;33(1):11-4. doi: 10.1016/j.joen.2006.09.005. PMID 17185119
- [Background] Al-Rawhani AH, Gawdat SI, Wanees Amin SA. Effect of Diclofenac Potassium Premedication on Postendodontic Pain in Mandibular Molars with Symptomatic Irreversible Pulpitis: A Randomized Placebo-Controlled Double-Blind Trial. J Endod. 2020 Aug;46(8):1023-1031. doi: 10.1016/j.joen.2020.05.008. Epub 2020 May 26. PMID 32470370